CLINICAL TRIAL: NCT02698215
Title: Combining Varenicline and Naltrexone for Smoking Cessation and Drinking Reduction
Brief Title: Combining Varenicline and Naltrexone for Smoking Cessation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Lara Ray, PhD, Associate Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VAR-NTX; R01DA041226 (NIH)
Record Dates: First submitted 2016-02-19; First posted 2016-03-03 (Estimated); Results first posted 2021-06-15 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-05

CONDITIONS: Nicotine Dependence; Alcohol Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder; Alcoholism | interventions — Varenicline; Naltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Varenicline plus Naltrexone (Experimental): VAR (1 mg twice daily) + NTX (50 mg once daily)
  Interventions: Drug: Varenicline plus Naltrexone
- Varenicline (Placebo Comparator): VAR (1 mg twice daily)
  Interventions: Drug: Varenicline

INTERVENTIONS:
Drug: Varenicline — Varenicline 1 mg twice daily
  Other Names: Chantix
  Arms: Varenicline
Drug: Varenicline plus Naltrexone — Varenicline 1 mg twice daily plus Naltrexone 50 mg once daily
  Other Names: Chantix; Revia
  Arms: Varenicline plus Naltrexone

SUMMARY:
This study is a double-blind, randomized clinical trial using a two group medication design consisting of the combination of VAR (1 mg twice daily) + NTX (50 mg once daily) and VAR (1 mg twice daily) + PLA (matched to NTX), for smoking cessation in a sample of heavy drinking daily smokers who want to quit smoking and reduce drinking.

DETAILED DESCRIPTION:
This study is a double-blind, randomized clinical trial using a two group medication design consisting of the combination of VAR (1 mg twice daily) + NTX (50 mg once daily) and VAR (1 mg twice daily) + PLA (matched to NTX), for smoking cessation in a sample of heavy drinking daily smokers who want to quit smoking and reduce drinking. All participants will be daily smokers (≥ 5 cig/day) who are also heavy drinkers according to the National Institute on Alcohol Abuse and Alcoholism (NIAAA) guidelines: for men, > 14 drinks per week or ≥ 5 drinks per occasion at least once per month over the past 12 months; for women, > 7 drinks per week or ≥ 4 drinks per occasion at least once per month over the past 12 months. A total of 274 participants will be randomized, 137 to each medication group.

ELIGIBILITY:
Inclusion Criteria:

1. Be treatment-seeking for smoking cessation and have a desire to reduce or quit drinking
2. Be between the ages of 21 and 65
3. Be able to provide informed consent
4. Smoke 5 or more cigarettes per day for the past year
5. Currently drink heavily according to the National Institute on Alcohol Abuse and Alcoholism (NIAAA) guidelines: for men, > 14 drinks per week or ≥ 5 drinks per occasion at least once per month over the past 12 months; for women, > 7 drinks per week or ≥ 4 drinks per occasion at least once per month over the past 12 months
6. Pass the physical exam and associated laboratory tests, as determined by study physician

Exclusion Criteria:

1. Have clinically significant alcohol withdrawal, indicated by a score ≥ 10 on the Clinical Institute Withdrawal Assessment for Alcohol (CIWA-Ar) and assessed at the in-person screening visits
2. Have lifetime DSM-V diagnosis of schizophrenia, bipolar disorder, a psychotic disorder, or any other psychiatric disorder as determined by the clinical interview
3. Have major depressive disorder within the past year requiring treatment as determined by the clinical interview using DSM-V criteria
4. Have a current or lifetime DSM-V diagnosis of a substance use disorder, other than for alcohol or nicotine, as determined by the clinical interview
5. Have a prior history of taking FDA approved medications (i.e. varenicline or bupropion) for smoking cessation
6. Be currently using any forms of nicotine replacement therapy (past use is acceptable)
7. Be currently using tobacco products other than cigarettes (such as e-cigarettes, cigars, or chewing tobacco)
8. Have a serious medical illness (significant cardiovascular disease; uncontrolled hypertension; hepatic or renal disease) that would contraindicate participation, as determined by the study physician
9. Be currently taking insulin or oral hypoglycemic medication
10. Be currently taking opioid pain medications or any form of opioid agonist maintenance therapy (such as methadone or buprenorphine)
11. Be currently taking any other psychoactive medications; such as anti-depressants, mood stabilizers, anti-seizure medications, sedatives-hypnotics, anxiolytics, stimulants or antipsychotics
12. Have self-reported use of cocaine, methamphetamine, heroin or other illicit drugs in the previous 60 days, verified by urine toxicology screen
13. For women, must not be pregnant (as indicated by self-report or a positive pregnancy test at any study visit), nursing, or planning to become pregnant while taking part in the study, and must agree to a reliable method of birth control

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lara Ray, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Addictions Laboratory, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Green R, Montoya AK, Ray LA. The relationship between drinking and smoking in a clinical trial for smoking cessation and drinking reduction. Exp Clin Psychopharmacol. 2022 Dec;30(6):873-883. doi: 10.1037/pha0000536. Epub 2021 Dec 30. PMID 34968106
- [Derived] Ray LA, Green R, Enders C, Leventhal AM, Grodin EN, Li G, Lim A, Hartwell E, Venegas A, Meredith L, Nieto SJ, Shoptaw S, Ho D, Miotto K. Efficacy of Combining Varenicline and Naltrexone for Smoking Cessation and Drinking Reduction: A Randomized Clinical Trial. Am J Psychiatry. 2021 Sep 1;178(9):818-828. doi: 10.1176/appi.ajp.2020.20070993. Epub 2021 Jun 3. PMID 34080890

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Varenicline Plus Naltrexone | Varenicline
Started | 83 | 82
Completed | 55 | 64
Not Completed | 28 | 18

BASELINE CHARACTERISTICS:
Population: 1 participant is missing data from the Cotinine and Alcohol Use Disorder (AUD) Severity baseline characteristics.
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline Plus Naltrexone | Varenicline | Total
Number analyzed (Participants) | 83 | 82 | 165
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.24 (12.42) | 42.07 (11.75) | 41.55 (12.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 32 | 63
  Male | 52 | 50 | 102
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 13 | 25
  Not Hispanic or Latino | 71 | 69 | 140
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 40 | 36 | 76
  White | 27 | 29 | 56
  More than one race | 5 | 7 | 12
  Unknown or Not Reported | 4 | 8 | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 83 | 82 | 165
Smoking Days (Timeline Followback) [Mean (Standard Deviation); unit: days] — Timeline Followback (TLFB) is a calendar-assisted interview where participants report the number of cigarettes they consumed over a specified assessment period. Participcants were asked to report whether they consumed a cigarette in the 30 days prior to the baseline visit. Smoking Days is the sum of days participants reported smoking a cigarette in the 30 days prior to the baseline visit.
  days | 28.94 (3.37) | 29.39 (1.49) | 29.16 (2.61)
Cigarettes per Smoking Day (Timeline Followback) [Mean (Standard Deviation); unit: cigarettes] | 14.21 (8.39) | 14.10 (7.79) | 14.16 (8.07)
Expired Alveolar CO Level (ppm) [Mean (Standard Deviation); unit: ppm] | 11.65 (6.25) | 9.68 (7.34) | 10.67 (6.86)
Urine Cotinine Levels (ng/ml) [Mean (Standard Deviation); unit: ng/ml] — Cotinine was assessed using a urine cotinine test (NicAlertTM), a rapid test utilizing semiquantitative immunoassay technology to detect tobacco from cigarettes with a score of 3 or higher (100-200ng/mL) indicating recent tobacco exposure.
  ng/ml | 5.50 (1.14) | 5.37 (1.05) | 5.44 (1.09)
Fagerstrom Test for Nicotine Dependence (FTND) Score [Mean (Standard Deviation); unit: units on a scale] — Fagerstrom Test for Nicotine Dependence (FTND) score is a self-report measure used to assess for severity of nicotine dependence. It consists of 6 items, with 2 items rated on a 4-point Likert scale (0 = less severe response, 3 = more severe response) and 4 items rated on a 2-point Likert scale (0 = less severe response, 1 = more severe response). A summary score (range: 0 - 10) is used to indicate severiety of nicotine dependence with greater scores indicating more severe nicotine dependence.
  units on a scale | 4.64 (2.26) | 4.61 (2.35) | 4.63 (2.30)
Drinking Days (Timeline Followback) [Mean (Standard Deviation); unit: days] — Timeline Followback (TLFB) is a calendar-assisted interview where participants report how much alcohol they consumed over a specified assessment period. Participcants were asked to report whether they consumed any alcohol on each calendar day in the 30 days prior to the baseline visit. Drinking Days is the sum of days participants reported consuming any alcohol in the 30 days prior to the baseline visit.
  days | 20.71 (8.08) | 19.63 (7.92) | 20.17 (8.00)
Drinks per Drinking Day (Timeline Followback) [Mean (Standard Deviation); unit: drinks per drinking day] | 6.50 (4.65) | 6.44 (3.76) | 6.47 (4.22)
Heavy Drinking Days (Timeline Followback) [Mean (Standard Deviation); unit: heavy drinking days] — Timeline Followback (TLFB) is a calendar-assisted interview where participants report how much alcohol they consumed over a specified assessment period. A trained interviewer records the number of standard drinks consumed on each day in the in the 30 days prior to the baseline visit. Heavy drinking was defined according to National Institute on Alcohol Abuse and Alcoholism (NIAAA) criteria of 4+ drinks/day for men and 3+ drinks/day for women. Heavy drinking days was defined as the number of days participants met criteria for heavy drinking in the 30 days prior to the baseline visit.
  heavy drinking days | 12.87 (9.55) | 12.30 (8.84) | 12.59 (9.18)
Alcohol Use Disorder Severity (Structured Clinical Interview for DSM-5) [Count of Participants; unit: Participants] — Population: One participant was missing DSM-5 AUD diagnosis data from the VAR+NTX group.
  Participants
    number analyzed (Participants) | 82 | 82 | 164
    None | 24 | 24 | 48
    Mild | 27 | 22 | 49
    Moderate | 19 | 23 | 42
    Severe | 12 | 13 | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Expired Carbon Monoxide Level <=5ppm
Description: Outcome for smoking cessation aim was Expired Carbon Monoxide level, which was used to determine whether a participant successfully abstained from cigarettes. 7 day point prevalence of nicotine abstinence was bioverified by Expired Carbon Monoxide reading of <= 5ppm at the 26-week follow-up visit.
Time Frame: 26 weeks post-quit
Population: Intent to Treat.
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline Plus Naltrexone | Varenicline
Number analyzed (Participants) | 83 | 82
Participants | 22 | 37

2. Secondary Outcome: Drinks Per Drinking Day
Description: Outcome for drinking reduction aim - Number of Drinks per Drinking Day
Time Frame: 26 weeks post-quit
Population: Intent to Treat
Measure: Mean (Standard Error); unit: drinks per drinking day
Arm/Group | Varenicline Plus Naltrexone | Varenicline
Number analyzed (Participants) | 83 | 82
drinks per drinking day | 3.1242 (1.0281) | 3.5121 (.9594)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected at each in-person visit (6 visits) during the medication period (approximately 12 weeks or 3 months).
Arm/Group | Varenicline Plus Naltrexone | Varenicline
All-Cause Mortality (participants affected / at risk) | 0/83 | 0/82
Serious Adverse Events (participants affected / at risk) | 0/83 | 0/82
Other Adverse Events (participants affected / at risk) | 63/83 | 64/82
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline Plus Naltrexone (N=83) | Varenicline (N=82)
nausea (Gastrointestinal disorders) | 38 (39) | 28 (29)
vomiting (Gastrointestinal disorders) | 8 (9) | 11 (12)
constipation (Gastrointestinal disorders) | 5 (5) | 3 (4)
diarrhea (Gastrointestinal disorders) | 4 (4) | 3 (3)
upset stomach (Gastrointestinal disorders) | 3 (4) | 8 (9)
decreased appetite (Gastrointestinal disorders) | 4 (4) | 0 (0)
increased appetite (Gastrointestinal disorders) | 1 (1) | 0 (0)
decreased bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0)
acid reflux (Gastrointestinal disorders) | 0 (0) | 1 (1)
headache (Nervous system disorders) | 15 (17) | 8 (10)
migraine (Nervous system disorders) | 1 (1) | 0 (0)
loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
dizziness (Nervous system disorders) | 1 (1) | 2 (2)
seizure (Nervous system disorders) | 0 (0) | 1 (1)
depression (Psychiatric disorders) | 6 (6) | 1 (1)
abnormal dreams (Psychiatric disorders) | 13 (13) | 17 (18)
anxiety (Psychiatric disorders) | 3 (3) | 3 (3)
mood swings (Psychiatric disorders) | 1 (1) | 0 (0)
dry mouth (Endocrine disorders) | 3 (3) | 2 (2)
low blood sugar (Endocrine disorders) | 0 (0) | 1 (1)
borderline diabetes (Endocrine disorders) | 1 (1) | 0 (0)
hyperglycemia (Endocrine disorders) | 1 (1) | 0 (0)
earache (Ear and labyrinth disorders) | 0 (0) | 1 (1)
ear infection (Ear and labyrinth disorders) | 1 (1) | 1 (1)
tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
bloody nose (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
sinus infection (Infections and infestations) | 1 (1) | 0 (0)
flu (Infections and infestations) | 2 (2) | 5 (5)
cold (Infections and infestations) | 4 (4) | 12 (12)
respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
fever (Infections and infestations) | 1 (1) | 3 (3)
runny nose (Infections and infestations) | 0 (0) | 1 (1)
elevated blood pressure (Cardiac disorders) | 1 (1) | 1 (1)
cardiac event (Cardiac disorders) | 1 (1) | 1 (1)
rapid heartbeat (Cardiac disorders) | 2 (2) | 0 (0)
difficulty breathing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
chest discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
sweating (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
skin irritation (Skin and subcutaneous tissue disorders) | 5 (8) | 9 (11)
joint pain or swelling (Musculoskeletal and connective tissue disorders) | 7 (8) | 5 (6)
fractured ribs (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
dental pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
mouth pain from wisdom tooth growth (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
hypersensitivity in teeth and mouth (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0)
neon green urine (Renal and urinary disorders) | 2 (2) | 0 (0)
pink eye (Eye disorders) | 1 (1) | 0 (0)
eye twitch (Eye disorders) | 0 (0) | 1 (1)
light sensitivity (Eye disorders) | 0 (0) | 1 (1)
uterine biopsy procedure (Reproductive system and breast disorders) | 1 (1) | 0 (0)
bartholin duct cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
yeast infection (Reproductive system and breast disorders) | 0 (0) | 2 (4)
feeling high (General disorders) | 0 (0) | 1 (1)
dehydration (General disorders) | 1 (1) | 1 (1)
extra thirsty (General disorders) | 0 (0) | 1 (1)
hair loss (General disorders) | 0 (0) | 1 (1)
decreased sex drive (General disorders) | 1 (1) | 1 (1)
weight gain (General disorders) | 0 (0) | 1 (1)
metallic taste (General disorders) | 1 (1) | 0 (0)
elevated cholesterol (General disorders) | 0 (0) | 1 (1)
decreased concentration (General disorders) | 1 (1) | 0 (0)
tired (General disorders) | 10 (10) | 3 (3)
fatigue (General disorders) | 4 (4) | 5 (5)
apathetic (General disorders) | 2 (2) | 1 (1)
trouble sleeping (General disorders) | 7 (9) | 5 (5)
confusion (General disorders) | 1 (1) | 0 (0)
irritability (General disorders) | 6 (6) | 10 (11)
jittery or shaky (General disorders) | 4 (4) | 2 (2)
tension (General disorders) | 0 (0) | 1 (1)
hot flashes (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-04-01): https://cdn.clinicaltrials.gov/large-docs/15/NCT02698215/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/15/NCT02698215/SAP_001.pdf